CLINICAL TRIAL: NCT03159871
Title: Closing Uterine Incision During C-section Using Barbed Suture (Stratafix) or Vicryl Suture: a Randomized Control Study
Brief Title: Closing Uterine Incision During C-section Using Barbed Suture (Stratafix) or Vicryl Suture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, Leon Grin, Gynecological Doctor, Barzilai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: BRZ 0018-16 CTIL
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Cesarean Section
Keywords: Cesarean section; C- section; Suture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stratafix suture (Experimental)
  Interventions: Device: Stratafix suture
- Vicryl suture (Active Comparator)
  Interventions: Device: Vicryl suture

INTERVENTIONS:
Device: Stratafix suture — Stratafix barbed sutures during C-Sections.
  Arms: Stratafix suture
Device: Vicryl suture — Standart Vicryl suture during C- Sections.
  Arms: Vicryl suture

SUMMARY:
A Randomized prospective single blinded trial. The investigator seek to evaluate the surgical outcome of Stratafix barbed suture compared to standart Vicryl sutures in reducing the suturing time during C-Section.

DETAILED DESCRIPTION:
A Randomized prospective single blinded trial. The investigator seek to evaluate the surgical outcome of Stratafix barbed suture compared to standart Vicryl sutures in reducing the suturing time during C-Section. In addition, the need of additional sutures to control bleeding after the 2- layer closure will be estimated.These will be the primary outcome measures. The secondary outcome measures will be factors related to the blood loss at the time of the uterine closure, surgical complications, duration of hospital stay, postoperative infection (endometritis) and wound infection..

ELIGIBILITY:
Inclusion Criteria:

• Pregnant patients with an obstetrical indication for delivery by Cesarean section

Exclusion Criteria:

• Patients with blood clotting disorders.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females
Enrollment: 73 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-24 (Actual)

PRIMARY OUTCOMES:
Time required for uterine closure. | From the beginning of first uterine suture till the last suture ending uterine incision complete closure and any additional hemostatic sutures if applicable. The estimated period of time is 8 minutes (average).
  Time measured in minutes and seconds

SECONDARY OUTCOMES:
Blood loss during uterine closure | Estimated period of time is 4 days.
  Intraoperative during uterine closure and by blood work during post-operative hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Barzilai Medical Center, Ashkelon, Israel

REFERENCES:
- [Background] Greenberg JA, Goldman RH. Barbed suture: a review of the technology and clinical uses in obstetrics and gynecology. Rev Obstet Gynecol. 2013;6(3-4):107-15. PMID 24920976
- [Background] Giampaolino P, De Rosa N, Tommaselli GA, Santangelo F, Nappi C, Sansone A, Bifulco G. Comparison of bidirectional barbed suture Stratafix and conventional suture with intracorporeal knots in laparoscopic myomectomy by office transvaginal hydrolaparoscopic follow-up: a preliminary report. Eur J Obstet Gynecol Reprod Biol. 2015 Dec;195:146-150. doi: 10.1016/j.ejogrb.2015.10.011. Epub 2015 Oct 24. PMID 26540594